CLINICAL TRIAL: NCT06998615
Title: Correlation Between Shoulder Impingement and Cervical Proprioception
Acronym: CP
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mustafa Yahia Abdelaziz Ebrahim Basha, principle investigator : mostafa yahia abdelaziz ibrahim, Cairo University
Other Study IDs: P.T.REC/012/005804
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Shoulder Impingement
Keywords: shoulder impingement; neck proprioception; correlation; cervical proprioception
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- shoulder impingement group: thirty four subjects with shoulder impingement will be included in this group
  Interventions: Other: shoulder impingement group
- normal subjets: thirty four normal subjects will be included in this group
  Interventions: Other: normal subjects

INTERVENTIONS:
Other: shoulder impingement group — the Patients with shoulder impingement syndrome in this group had at least 3 out of the following 6 criteria 1) positive "Neer's sign"; 2) positive "Hawkins' sign"; 3) pain on active shoulder elevation in the scapular plane, 4) pain on the C5-C6 dermatome; 5) pain on palpation of the rotator cuff tendons and 6) pain with resisted isometric abduction.
  Groups: shoulder impingement group
Other: normal subjects — the subjects in this group had no pain or disability in shoulder
  Groups: normal subjets

SUMMARY:
this study will be conducted to evaluate the correlation between shoulder impingement and cervical proprioception

DETAILED DESCRIPTION:
Shoulder pain is one of the most common complaints in musculoskeletal practice, whether it comes from impingement syndrome or a defect in rotator cuff muscles .Shoulder pain is considered to be the third most common complaint in musculoskeletal practice, with a prevalence of 7% to 34% .Shoulder impingement is a syndrome where there is entrapment of soft tissue through the shoulder joint, with a prevalence of 44% to 65% of all shoulder complaints. Shoulder impingement has multiple causes, whether functional, degenerative, and anatomical and mechanical causes .Shoulder impingement classified to primary and secondary. Secondary impingement is subdivided into internal and external impingement .Proprioception components are joint position sense, kinesthesia, sense of force, sense of change of velocity. joint position sense is our perception of position of the joint or limb it divided to active/passive joint position sense, it means that the person can relocate the position of the joint or the limb to the same position after the joint or limb is moved.the muscle receptor helping in identifying the limb position and movement through changeling in neural signaling in the sensory receptor, giving the neurological control and basis of proprioception to sensory receptors located in the skin, muscles, and joints, so the proprioception is considered to be a loop of feedforward and feedback signals between sensory receptor and the nervous system. sixty eight subjects with shoulder impingement syndrome will be joined to this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Patients diagnosed with shoulder impingement
* Age: Patients aged between 25 and 45 years.
* Pain and mobility issues: Patients must report mild to moderate pain and/or restricted range of motion (ROM) in shoulder joint .
* Ability to provide informed consent: Participants must be able to understand the study protocol and provide written informed consent to participate.
* Medical stability: Patients must be medically stable and able to engage in physical assessment

Exclusion Criteria:

* any patient aged below 25 or above 45 years old
* Subjects have malignancy: Patients with severe neurological, musculoskeletal, disorders that could interfere with the study interventions
* Subjects have history of shoulder trauma, fractures and surgeries:
* Subjects have neck dysfunction
* Cognitive impairment: Patients with significant cognitive impairment or mental health conditions that would hinder their ability to understand or comply with the study protocol.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: sixty eight subjects will be included in this study; thirty four with shoulder impingement syndrome and thirty four healthy subjects with no shoulder impingement
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
joint position error (cervical proprioception) | up to thirty minutes
  neck proprioception by Joint Position Error (JPE) using LASER beam Point tool and it's conducted as patient sitting 90 cm away from the target map on the wall ad a light weight headband with laser pointer is placed on the patient head, the patient is asked to focus on the center of the map while eye open then the patient asked to close his eyes and move his head in one plane and back to the starting point as accurately as possible and indicate verbally that he back to the starting position before opening his eyes, he repeated for 6 times in each plane and the distance between the starting point and the ending point is measured and then converted to degrees the patient is diagnosed to has a proprioception deficit if the mean error of any direction in more than 4.5 degrees
shoulder disablity | up to thirty minutes
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use.he pain scale is summed up to a total of 50 while the disability scale sums up to 80. The total SPADI score is expressed as a percentage. A score of 0 indicates best 100 indicates worst.
pain intensity | up to thirty minutes
  Pain will be assed with numerical analog scale (NPRS) in which a respondent selects a whole number (0-10 cm) that best reflects the intensity of his/her pain. 0 mean no pain and 10 mean maximum pain